CLINICAL TRIAL: NCT00086554
Title: Procurement of Clinical Specimens for Immunologic or Genetic Studies in Inflammatory Bowel Diseases
Brief Title: Collection of Specimens for Study of Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040231; 04-I-0231
Record Dates: First submitted 2004-07-02; First posted 2004-07-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-01-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Surgery; Intestinal Resection; Blood Sample
MeSH Terms: conditions — Inflammatory Bowel Diseases

SUMMARY:
This study will collect tissue specimens to be used for research on inflammatory bowel disease. The tissues will be used to explore why people get inflammatory bowel disease and to try to develop new treatments based on the study results. Tissue from patients with IBD will be compared with that from patients who do not have the disease

Patients who undergo bowel surgery for inflammatory bowel disease (IBD) or another bowel disorder may be eligible for this study. Patients with IBD must be at least 4 years of age; those with another disorder must be 18 years of age or older.

Participants undergo bowel surgery for their disease. Some of the intestinal tissue removed during the surgery that is not needed for medical care, such as for pathological examination, is provided to researchers for study under this protocol. In addition, patients with IBD provide a blood sample for genetic testing. Several genetic variations, or mutations, may increase the risk of developing IBD; blood samples from patients may help identify these variations.

DETAILED DESCRIPTION:
Our ongoing natural history studies of the etiology and immune abnormalities of the group of diseases known collectively as the inflammatory bowel diseases require access to clinical samples of intestinal tissue as well as blood samples for genotyping. This protocol provides a mechanism for procurement of intestinal samples obtained at the time of medically-indicated surgical procedures from patients with IBD or some other non-IBD diagnosis (to act as a control group). In addition it allows for the procurement of blood for DNA preparation as more IBD susceptibility genes are discovered and we further our work on association of genetic polymorphisms/mutations with the phenotype and immune abnormalities observed in our IBD patients.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SUBJECTS WITH INFLAMMATORY BOWEL DISEASE:

  1. Presence of idiopathic inflammatory bowel disease as established by prior endoscopic, histologic, and/or radiographic findings.
  2. Ability to give consent or have legally authorized person give consent and agree to sample storage.

EXCLUSION CRITERIA FOR SUBJECTS WITH INFLAMMATORY BOWEL DISEASE:

1. Less than 4 years old.

INCLUSION CRITERIA FOR SUBJECTS WITHOUT INFLAMMATORY BOWEL DISEASE:

1. Absence of idiopathic inflammatory bowel disease as established by tests that exclude these diagnoses.
2. Ability to give consent and agree to sample storage.

EXCLUSION CRITERIA FOR SUBJECTS WITHOUT INFLAMMATORY BOWEL DISEASE:

1. Less than 18 years of age.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07-01; Study Completion 2010-01-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States